CLINICAL TRIAL: NCT03036592
Title: MTNR1B SNP*Food Timing Interaction on Glucose Control in a Late Eater Mediterranean Population
Brief Title: MTNR1B SNP*Food Timing Interaction on Glucose Control
Acronym: ONTIME-MT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, PROF. MARTA GARAULET AZA, Full Professor, Universidad de Murcia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2017ES00001
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Non-Diabetic Disorder of Endocrine Pancreas
Keywords: Glucose tolerance test, MTNR1B, nutrigenomics, food timing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Early OGTT, then late OGTT in MTNR1B CC (Experimental): Oral glucose tolerance test (OGTT) in homozygous non-carriers (CC) for MTNR1B rs10830963 in Early and Late conditions
  Interventions: Behavioral: Early OGTT; Behavioral: Late OGTT
- Early OGTT, then late OGTT in MTNR1B CG (Experimental): Oral glucose tolerance test (OGTT) in heterozygous (CG) risk allele carriers for MTNR1B rs10830963 in Early and Late conditions
  Interventions: Behavioral: Early OGTT; Behavioral: Late OGTT
- Early OGTT, then late OGTT in MTNR1B GG (Experimental): Oral glucose tolerance test (OGTT) in homozygous (GG) risk allele carriers for MTNR1B rs10830963 in Early and Late conditions
  Interventions: Behavioral: Early OGTT; Behavioral: Late OGTT
- Late OGTT, then Early OGTT in MTNR1B CC (Experimental): Oral glucose tolerance test (OGTT) in heterozygous (CG) risk allele carriers for MTNR1B rs10830963 in Early and Late conditions
  Interventions: Behavioral: Early OGTT; Behavioral: Late OGTT
- Late OGTT, then Early OGTT in MTNR1B CG (Experimental): Oral glucose tolerance test (OGTT) in heterozygous (CG) risk allele carriers for MTNR1B rs10830963 in Early and Late conditions
  Interventions: Behavioral: Early OGTT; Behavioral: Late OGTT
- Late OGTT, then Early OGTT in MTNR1B GG (Experimental): Oral glucose tolerance test (OGTT) in heterozygous (CG) risk allele carriers for MTNR1B rs10830963 in Early and Late conditions
  Interventions: Behavioral: Early OGTT; Behavioral: Late OGTT

INTERVENTIONS:
Behavioral: Early OGTT — Oral glucose tolerance test using identical mixed 75 gr of glucose under early condition (4 hours before habitual bedtime)
Behavioral: Late OGTT — Oral glucose tolerance test using identical mixed 75 gr of glucose under late condition (1 hour before habitual bedtime)

SUMMARY:
The purpose of this investigation is to assess the role of melatonin receptor 1B (MTNR1B) single nucleotide polymorphism (SNP)*food timing interaction on glucose control in the deleterious effect in a vulnerable population with regular exposure to concurrent high melatonin and food intake as late night eaters (those having dinner within 2.5 h before their usual bed time). With the results from this study, we expect to advance our understanding of the role of endogenous melatonin on glucose metabolism in late night eaters and carriers of the MTNR1B risk allele, with potential implications on the guidelines to mitigate risk of type 2 diabetes in late night eaters and carriers of the MTNR1B risk allele.

DETAILED DESCRIPTION:
Late-night dinner eating is associated with increased risk for type-2-diabetes. The underlying mechanism is unclear. One explanatory hypothesis is that the concurrence of elevated circulating melatonin and high glucose concentrations (characterizing late-eating) leads to impaired glucose-tolerance. However, to date, no study has tested the influence of physiological melatonin concentrations on glucose tolerance. The discovery of melatonin receptor MTNR1B as a diabetes risk gene provides evidence for a role of physiological levels of melatonin in glucose control.

The aim of the current study is to test the hypothesis that the concurrence of meal timing with elevated endogenous melatonin concentrations results in impaired glucose control and that this effect is stronger in homozygous MTNR1B risk carriers than in non-carriers. To do so we will test glucose tolerance using identical mixed meals under two glucose oral tolerance test (OGTT) conditions: a) delayed OGTT or Late Eating (LE): starting1 hour before their usual bed time, b) advanced OGTT or Early Eating (EE): starting 4 hours before habitual bed time, in a randomized, cross-over study design.

These findings could support a clinical application for the screening of this SNP and the possibility of implementing tailored and cost-effective behavioral interventions to prevent type 2 diabetes in vulnerable populations.

These goals will be achieved through a specific approach:

• Interventional (randomized, cross-over controlled trials) (Aim 1): To study the potential interaction between meal timing (dinner) and genetic variants MTNR1B for glucose tolerance (n=1000).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index: > 18.5 o < 40 kg/m2
* Age: between 18 and 65 year of age
* European ancestry
* Day workers

Exclusion Criteria:

* Receiving treatment with thermogenic, lipogenic, or drugs
* Diabetes mellitus, chronic renal failure, hepatic diseases, or cancer diagnosis
* Bulimia diagnosis, prone to binge eating
* Undergoing treatment with Type 2 diabetes mellitus (high blood sugar) medications such as Metformin or other non-Metformin oral anti-diabetic drugs such as sulfonylureas, meglitinides, or glitazones
* Undergoing treatment with Corticosteroids/steroids, Growth hormone, Anticoagulant medicines, or blood thinners, Beta blockers for hypertension, Medications for sleep, Fluvoxamine, Opioids or Amphetamines, Tranquilizers, nonsteroidal anti-inflammatory drugs.
* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 889 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Purificación Gomez Abellan, PHD, Study Chair — Universidad de Murcia
Locations (1):
- University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garaulet M, Lopez-Minguez J, Dashti HS, Vetter C, Hernandez-Martinez AM, Perez-Ayala M, Baraza JC, Wang W, Florez JC, Scheer FAJL, Saxena R. Interplay of Dinner Timing and MTNR1B Type 2 Diabetes Risk Variant on Glucose Tolerance and Insulin Secretion: A Randomized Crossover Trial. Diabetes Care. 2022 Mar 1;45(3):512-519. doi: 10.2337/dc21-1314. PMID 35015083

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1457 patients were recruited from January 2017 to March 2020.
Pre-assignment Details: 845 of 1457 participants were included in this study. Of those not included, 200 declined to participate, 176 did not meet inclusion criteria, 192 lost to follow-up and 44 did not have the complete data. Nevertheless, because the genotype was not known until finishing recruitment, we cannot add the information in each arm of the started, etc.
Groups:
- Early OGTT, Then Late OGTT in MTNR1B CC: Oral glucose tolerance test (OGTT) in homozygous non-carriers (CC) for MTNR1B rs10830963 in Early condition. After a washout period of 1 week, OGTT was performed in Late condition in a randomized cross-over study design.
  Early OGTT: Oral glucose tolerance test using identical mixed 75 gr of glucose under early condition (4 hours before habitual bedtime)
  Late OGTT: Oral glucose tolerance test using identical mixed 75 gr of glucose under late condition (1 hour before habitual bedtime)
- Early OGTT, Then Late OGTT in MTNR1B CG: Oral glucose tolerance test (OGTT) in heterozygous (CG) risk allele carriers for MTNR1B rs10830963 in Early condition. After a washout period of 1 week, OGTT was performed in Late condition in a randomized cross-over study design.
  Early OGTT: Oral glucose tolerance test using identical mixed 75 gr of glucose under early condition (4 hours before habitual bedtime)
  Late OGTT: Oral glucose tolerance test using identical mixed 75 gr of glucose under late condition (1 hour before habitual bedtime)
- Early OGTT, Then Late OGTT in MTNR1B GG: Oral glucose tolerance test (OGTT) in homozygous (GG) risk allele carriers for MTNR1B rs10830963 in Early condition. After a washout period of 1 week, OGTT was performed in Late condition in a randomized cross-over study design.
  Early OGTT: Oral glucose tolerance test using identical mixed 75 gr of glucose under early condition (4 hours before habitual bedtime)
  Late OGTT: Oral glucose tolerance test using identical mixed 75 gr of glucose under late condition (1 hour before habitual bedtime)
- Late OGTT, Then Early OGTT in MTNR1B CC: Oral glucose tolerance test (OGTT) in homozygous (GG) risk allele carriers for MTNR1B rs10830963 in Late condition. After a washout period of 1 week, OGTT was performed in Early condition in a randomized cross-over study design.
  Late OGTT: Oral glucose tolerance test using identical mixed 75 gr of glucose under late condition (1 hour before habitual bedtime)
  Early OGTT: Oral glucose tolerance test using identical mixed 75 gr of glucose under early condition (4 hours before habitual bedtime)
- Late OGTT, Then Early OGTT in MTNR1B CG: Oral glucose tolerance test (OGTT) in heterozygous (CG) risk allele carriers for MTNR1B rs10830963 in Late condition. After a washout period of 1 week, OGTT was performed in Early condition in a randomized cross-over study design.
  Late OGTT: Oral glucose tolerance test using identical mixed 75 gr of glucose under late condition (1 hour before habitual bedtime)
  Early OGTT: Oral glucose tolerance test using identical mixed 75 gr of glucose under early condition (4 hours before habitual bedtime)
- Late OGTT, Then Early OGTT in MTNR1B GG: Oral glucose tolerance test (OGTT) in homozygous (GG) risk allele carriers for MTNR1B rs10830963 in Late condition. After a washout period of 1 week, OGTT was performed in Early condition in a randomized cross-over study design.
  Late OGTT: Oral glucose tolerance test using identical mixed 75 gr of glucose under late condition (1 hour before habitual bedtime)
Period: First Visit (1day)
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Started | 221 | 193 | 36 | 202 | 149 | 44
Completed | 221 | 193 | 36 | 202 | 149 | 44
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (1week)
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Started | 221 | 193 | 36 | 202 | 149 | 44
Completed | 221 | 193 | 36 | 202 | 149 | 44
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Visit (1day)
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Started | 221 | 193 | 36 | 202 | 149 | 44
Completed | 221 | 193 | 36 | 202 | 149 | 44
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Early OGTT, Then Late OGTT in MTNR1B CC: Oral glucose tolerance test (OGTT) in homozygous non-carriers (CC) for MTNR1B rs10830963 in Early condition. After a washout period of 1 week, OGTT was performed in Late condition in a randomized cross-over study design.
- Early OGTT, Then Late OGTT in MTNR1B CG: Oral glucose tolerance test (OGTT) in heterozygous (CG) risk allele carriers for MTNR1B rs10830963 in Early condition. After a washout period of 1 week, OGTT was performed in Late condition in a randomized cross-over study design.
- Early OGTT, Then Late OGTT in MTNR1B GG: Oral glucose tolerance test (OGTT) in homozygous (GG) risk allele carriers for MTNR1B rs10830963 in Early condition. After a washout period of 1 week, OGTT was performed in Late condition in a randomized cross-over study design.
- Late OGTT, Then Early OGTT in MTNR1B CC: Oral glucose tolerance test (OGTT) in homozygous non-carriers (CC) for MTNR1B rs10830963 in Late condition. After a washout period of 1 week, OGTT was performed in Early condition in a randomized cross-over study design.
- Late OGTT, Then Early OGTT in MTNR1B CG: Oral glucose tolerance test (OGTT) in heterozygous (CG) risk allele carriers for MTNR1B rs10830963 in Late condition. After a washout period of 1 week, OGTT was performed in Early condition in a randomized cross-over study design.
- Late OGTT, Then Early OGTT in MTNR1B GG: Oral glucose tolerance test (OGTT) in homozygous (GG) risk allele carriers for MTNR1B rs10830963 in Late condition. After a washout period of 1 week, OGTT was performed in Early condition in a randomized cross-over study design.
- Total: Total of all reporting groups
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG | Total
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44 | 845
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (13) | 39 (14) | 36 (15) | 38 (14) | 39 (15) | 37 (16) | 38 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 136 | 30 | 143 | 107 | 32 | 600
  Male | 69 | 57 | 6 | 59 | 42 | 12 | 245
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 221 | 193 | 36 | 202 | 149 | 44 | 845
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) Glucose
Description: Glucose levels are measured along 120 minutes corresponding to at early and late condition in each visit. The Area Under the Curve was calculated as the sum of the area of several trapezoids. This trapezoids was obtained at times 0-30 min, 30-60 min, 60-90 min, 90-120 min. The values are the difference between the late and the early condition.
Time Frame: Along 120 minutes in visits 1 and 2
Measure: Mean (Standard Deviation); unit: mg*h/dL
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
mg*h/dL
  AUC_Glucose_EE (Early Eating) | 278.84 (49.12) | 268.92 (48.69) | 260.66 (45.30) | 282.21 (54.89) | 274.91 (55.55) | 282.19 (56.56)
  AUC_Glucose_LE (Late Eating) | 291.58 (49.73) | 300.51 (54.60) | 300.61 (61.35) | 300.70 (56.88) | 299.09 (57.74) | 320.32 (63.95)

2. Primary Outcome: Disposition Index (DI)
Description: Disposition Index (DI) is the product of insulin sensitivity times by the amount of insulin secreted in response to blood glucose levels. Disposition index is used as a measure of beta cell function and the ability of the body to dispose of a glucose load. This index was determined by this formula:
  DI= CIR × ISI, where CIR is the measure Corrected Insulin Response, and ISI is Insulin Sensitivity Index. The values are the difference between the late and the early condition.
  Higher DI indicates an increased beta cell function and increased ability of the body to dispose of a glucose load.
Time Frame: Along 120 minutes in visits 1 and 2
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
Index
  DI_EE | 3.44 (3.03) | 4.59 (6.42) | 5.04 (6.14) | 3.54 (3.04) | 3.83 (3.84) | 3.96 (3.61)
  DI_LE | 3.33 (3.66) | 2.97 (2.55) | 2.78 (1.67) | 3.19 (3.34) | 3.19 (2.50) | 3.04 (4.46)

3. Secondary Outcome: Corrected Insulin Response (CIR)
Description: The measure of Corrected Insulin Response (CIR) uses the insulin and glucose levels at minute 30, integrating these values in the formula:
  CIR= l30/(G30 × (G30 - 70)).The values are the difference between the late and the early conditions.
  CIR is an index that assesses the insulin secretion capacity of B cells. A low CIR implies hyposecretion in response to glucose levels.
Time Frame: At minute 30 during the visit 1 and 2.
Measure: Mean (Standard Deviation); unit: Index
Groups:
- Late OGTT, Then Early OGTT in MTNR1B GG Late OGTT, Then Early OGTT in MTNR1B CG: Oral glucose tolerance test (OGTT) in homozygous (GG) risk allele carriers for MTNR1B rs10830963 in Late condition. After a washout period of 1 week, OGTT was performed in Early condition in a randomized cross-over study design.
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG Late OGTT, Then Early OGTT in MTNR1B CG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
Index
  CIR_EE | 0.57 (0.60) | 0.70 (1.10) | 0.94 (1.41) | 0.58 (0.52) | 0.59 (0.45) | 0.53 (0.38)
  CIR_LE | 0.50 (0.46) | 0.44 (0.38) | 0.46 (0.23) | 0.53 (0.60) | 0.51 (0.45) | 0.36 (0.28)

4. Secondary Outcome: Insulin Sensitivity Index (ISI)
Description: Insulin Sensitivity Index is a measurement which integrates fasting glucose and insulin concentrations (0 min) and the mean of the glucose and insulin levels from 0 to 120 minutes (0, 30, 60, 90 and 120 min), from an OGTT, to measure insulin sensitivity. This formula allows its use in clinical settings as well as in large epidemiological studies. The values are the difference between the late and the early condition.
  Elevated ISI values typically indicate a favorable outcome. This index reflects the body's responsiveness to insulin, a hormone crucial for regulating blood sugar levels. Higher sensitivity to insulin suggests that cells efficiently utilize insulin's signals, promoting better blood sugar management. Lower ISI may lead to challenges in maintaining stable blood glucose levels and is often associated with conditions such as type 2 diabetes and metabolic syndrome.
Time Frame: Along 120min in visits 1 and 2
Measure: Mean (Standard Deviation); unit: Index
Groups:
- Early OGTT, Then Late OGTT in MTNR1B CC: Oral glucose tolerance test (OGTT) in homozygous non-carriers (CC) for MTNR1B rs10830963 in Early condition. After a washout period of 1 week, OGTT was performed in Late condition in a randomized cross-over study design.
  Early OGTT: Test glucose tolerance using identical mixed 75 gr of glucose under early condition (4 hours before habitual bedtime)
  Late OGTT: Test glucose tolerance using identical mixed 75 gr of glucose under late condition (1 hour before habitual bedtime)
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
Index
  ISI_EE | 7.36 (5.40) | 7.26 (4.38) | 6.42 (3.43) | 7.19 (5.02) | 7.40 (5.13) | 7.61 (3.91)
  ISI_LE | 8.11 (6.98) | 8.11 (6.34) | 7.32 (4.20) | 6.99 (4.91) | 7.59 (5.22) | 8.00 (6.66)

5. Secondary Outcome: Fasting Glucose
Description: Fasting glucose (or basal glucose) is a simple measurement of glucose concentrations at minute 0 to see how glucose levels rise immediately after an OGTT. The values are the difference between the late and the early condition.
Time Frame: At minute 0 in visit 1 and 2.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 212 | 193 | 36 | 202 | 149 | 44
mg/dL
  Fasting glucose_EE | 85.25 (7.73) | 84.36 (7.25) | 84.05 (5.75) | 84.37 (6.84) | 84.69 (7.71) | 83.01 (4.90)
  Fasting glucose_LE | 84.09 (7.15) | 84.92 (7.07) | 85.70 (6.90) | 84.70 (7.74) | 85.53 (6.8) | 83.87 (7.51)

6. Secondary Outcome: Fasting Insulin
Description: Fasting insulin (or basal insulin) is a simple measurement of insulin concentrations at minute 0 to see how insulin levels rise immediately after an OGTT.The values are the difference between the late and the early condition.
Time Frame: At minute 0 in visit 1 and 2
Measure: Mean (Standard Deviation); unit: µU/mL
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
µU/mL
  Fasting insulin_EE | 6.70 (4.51) | 6.30 (4.28) | 6.88 (3.73) | 6.67 (4.73) | 6.16 (3.58) | 5.63 (3.69)
  Fasting insulin_LE | 6.13 (4.48) | 5.70 (3.65) | 5.71 (2.73) | 6.50 (4.56) | 6.09 (3.83) | 5.52 (3.32)

7. Secondary Outcome: Serum Melatonin
Description: Measurement of serum melatonin is made at time 0 and at time 120 in both the early and late conditions of everyone.
Time Frame: At baseline and 120 minutes in visit 1 and 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 158 | 136 | 23 | 136 | 104 | 31
pg/mL
  Melatonin_t0_EE | 20.86 (12.32) | 19.50 (9.82) | 20.25 (10.70) | 19.20 (10.39) | 19.01 (10.87) | 23.13 (14.92)
  Melatonin_t120_EE | 25.81 (17.69) | 26.85 (22.10) | 25.72 (19.65) | 25.40 (18.03) | 21.83 (13.47) | 29.61 (26.63)
  Melatonin_t0_LE | 52.69 (40.34) | 53.16 (43.69) | 54.24 (35.21) | 49.32 (34.39) | 47.16 (41.14) | 55.33 (32.39)
  Melatonin_t120_LE | 79.36 (52.24) | 83.92 (60.28) | 93.83 (63.71) | 81.07 (55.86) | 74.06 (55.72) | 83.80 (44.87)

8. Secondary Outcome: Dim Light Melatonin Onset (DLMO) at Early Condition Only
Description: This measurement shows the decimal time of the onset of melatonin in dim light conditions. In the case of DLMO, we only performed this measure at the early condition in order to get the analysis of melatonin during 5 hours (4 hours before the habitual bedtime and 1 hour later), as it is described in literature (DOI: 10.1002/oby.23749).
Time Frame: Melatonin measured every half hour for 5 hours at Early condition in all participants
Population: We only performed this measure at the early condition in each arm
Measure: Mean (Standard Deviation); unit: decimal hours
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 43 | 40 | 12 | 42 | 29 | 8
decimal hours | 22.42 (1.33) | 22.03 (1.06) | 22.41 (0.92) | 22.50 (1.38) | 22.08 (1.13) | 22.39 (1.40)

9. Other Pre Specified Outcome: Temperature Record (Mean Value 10hours Daytime)
Description: Measured using a temperature sensor which records the temperature during 7 days. We only determined it during the washout period (neither early nor late conditions).
Time Frame: For 1 week between visit 1 and 2
Measure: Mean (Standard Deviation); unit: centigrade degrees
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
centigrade degrees | 32.94 (0.98) | 32.95 (1.09) | 33.24 (0.94) | 33.05 (0.98) | 32.91 (0.93) | 33.02 (0.95)

10. Other Pre Specified Outcome: Activity Record (Mean Value 10hours Daytime)
Description: During the seven days of the study, individuals wore a wristwatch in their non-dominant hand, that integrates two sensors: a temperature sensor, and an accelerometer sensor that records physical activity and body position data (G Acceleration Data Logger UA-004-64; Onset Computer, Bourne, MA, USA). Activity was expressed as the change in degrees per minute (Δ°/min). We calculated the average activity value during the 10 consecutive hours of maximum values. We only determined it during the washout period (neither early nor late conditions).
Time Frame: For 1 week between visit 1 and 2
Measure: Mean (Standard Deviation); unit: changes in degrees/min (Δ°/min)
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
changes in degrees/min (Δ°/min) | 42.69 (8.51) | 51.61 (85.33) | 42.62 (6.46) | 41.73 (9.12) | 43.83 (8.06) | 44.30 (8.31)

11. Other Pre Specified Outcome: Light Exposure (Mean Value 10hours Daytime)
Description: Measured using a light sensor during 7 days. We only determined it during the washout period (neither early nor late conditions).
Time Frame: For 1 week between the visits 1 and 2
Measure: Mean (Standard Deviation); unit: Lux log
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
Lux log | 0.82 (0.24) | 0.83 (0.24) | 0.77 (0.27) | 0.81 (0.25) | 0.81 (0.25) | 0.88 (0.32)

12. Other Pre Specified Outcome: Sleep Duration
Description: Sleep duration will be computed from self-reported. We only determined it during the washout period (neither early nor late conditions).
Time Frame: For 1 week between visit 1 and 2
Measure: Mean (Standard Deviation); unit: decimal hours
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
decimal hours | 7.43 (0.75) | 7.52 (0.79) | 7.58 (0.70) | 7.56 (0.82) | 7.46 (0.88) | 7.51 (0.69)

13. Other Pre Specified Outcome: Total Energy Intake
Description: Total energy intake in kcal/day will be computed with a 7-day dietary log. We only determined it during the washout period (neither early nor late conditions).
Time Frame: For 1 week between visit 1 and 2
Measure: Mean (Standard Deviation); unit: Kcal/day
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
Kcal/day | 1563.64 (529.39) | 1548.29 (552.64) | 1666.25 (633.62) | 1555.96 (625.39) | 1619.23 (695.37) | 1753.18 (719.78)

14. Other Pre Specified Outcome: Dietary Composition
Description: Macronutrient and micronutrient intake will be computed from 7-days of self-reported 24-hr dietary recalls.
  Percentage Kcal respect to the Total Energy Intake. We only determined it during the washout period (neither early nor late conditions).
Time Frame: For 1 week between visit 1 and 2
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
percentage
  Fat | 34.85 (7.01) | 33.95 (7.37) | 36.04 (8.25) | 33.94 (7.83) | 34.90 (8.04) | 35.85 (8.49)
  Proteins | 17.52 (3.41) | 18.26 (3.94) | 18.02 (3.92) | 18.18 (3.95) | 18.24 (3.48) | 17.57 (3.65)
  Carbohydrates | 47.17 (7.66) | 47.75 (7.42) | 46.85 (7.38) | 47.82 (8.33) | 46.64 (8.49) | 46.68 (7.58)

15. Other Pre Specified Outcome: Dietary Intake Timing
Description: Food timing will be self-reported and averaged across 7-days of 24-hour dietary recalls. We only determined it during the washout period (neither early nor late conditions).
Time Frame: For 1 week between visit 1 and 2
Measure: Mean (Standard Deviation); unit: decimal hours
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
decimal hours
  Start breakfast | 8.72 (0.98) | 8.68 (0.87) | 8.80 (0.92) | 8.74 (0.92) | 8.68 (0.83) | 8.66 (0.96)
  Start lunch | 14.66 (0.49) | 14.72 (0.53) | 14.60 (0.42) | 14.70 (0.52) | 14.71 (0.48) | 14.50 (0.38)
  Start dinner | 21.66 (0.53) | 21.61 (0.65) | 21.64 (0.49) | 21.61 (0.56) | 21.67 (0.54) | 21.54 (0.56)

16. Other Pre Specified Outcome: Physical Activity
Description: Assessed using the International Physical Activity Questionnaire (IPAQ). This international questionnaire measures physical activity through the amount of energy expended carrying out physical activity i.e., Metabolic Units (MET) minutes a week. The higher the MET, the more amount of physical activity the individual performs. This allows us to classify low, moderate, or vigorous activity. 7 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of at least 3000 MET minutes a week. We only determined it during the washout period (neither early nor late conditions).
  Formula for computation of Met-minutes:
  * Walking MET-minutes/week = 3.3 * walking minutes * walking "days"
  * Moderate MET-minutes/week = 4.0 * moderate-intensity activity minutes * moderate days
  * Vigorous MET-minutes/week = 8.0 * vigorous-intensity activity minutes * vigorous-intensity days
Time Frame: During the week of washout
Measure: Mean (Standard Deviation); unit: Metabolic Units (MET)-minutes/week
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
Metabolic Units (MET)-minutes/week | 4066.98 (5898.97) | 4548.62 (5060.76) | 4560.41 (5779.47) | 4646.63 (4877.34) | 4429.64 (5284.58) | 4608.31 (4765.35)

17. Other Pre Specified Outcome: Chronotype
Description: Assessed using the Morningness-Eveningness Questionnaire (MEQ). Its main purpose is to measure whether a person's circadian rhythm produces peak alertness in the morning, in the evening, or in between. It is a score that indicates the degree to which the individual favors the morning over the night. We only determined it during the washout period (neither early nor late conditions).
  Values:
  Min: 17 Max: 86
  Explanation:
  17-30: extreme eveningness 31-41: eveningness 42-58: neither 59-69: morningness 70-86: extreme morningness
Time Frame: During the week of washout
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
score | 51.15 (9.42) | 51.75 (8.90) | 49.83 (10.70) | 51.35 (10.15) | 51.65 (10.32) | 51.11 (8.97)

18. Other Pre Specified Outcome: Emotional Eating
Description: Assessed using the Emotional Eating Questionnaire (EEQ). This questionnaire classifies individuals based on the relationship between food intake and emotions.
  Score between 0 and 30. We only determined it during the washout period (neither early nor late conditions).
  Explanation:
  0-5: nothing emotional 5-10: less emotional 10-20: emotional 20-30: Very emotional
Time Frame: During the week of washout
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
score | 11.10 (6.26) | 10.64 (5.74) | 11.16 (6.32) | 10.98 (6.16) | 10.81 (6.28) | 10.54 (5.79)

19. Other Pre Specified Outcome: Sleep Quality
Description: Assessed using the Pittsburgh Sleep Quality Index (PSQI). This questionnaire is used to quantitatively assess the quality of sleep. 7 scores are obtained that inform us about various aspects of sleep quality. We only determined it during the washout period (neither early nor late conditions).
  Score between 0 and 21. Total score of the questionnaire is divided into 7 items. Those items have a score from 0 (no problem) to 3 (severe problem).
  0-5: sleep quality optimum 6-21: sleep disorders
Time Frame: During the week of washout
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
score | 6.05 (3.05) | 6.15 (3.15) | 6.75 (3.25) | 7.00 (3.74) | 6.84 (3.36) | 6.49 (3.29)

20. Other Pre Specified Outcome: Insomnia
Description: Assessed using the Insomnia Severity Index (ISI). This questionnaire has 5 items and is used to assess the possible existence of sleep problems. According to the score obtained, a classification is made from no insomnia to severe clinical insomnia. We only determined it during the washout period (neither early nor late conditions).
  Score ranges between 0 and 28
  Explanation:
  0-7: no insomnia 8-14: subclinical insomnia 15-21: moderate insomnia 22-28: severe insomnia The higher the score, the more harmful
Time Frame: During the week of washout
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
score | 6.44 (4.83) | 6.63 (4.99) | 7.86 (5.48) | 7.04 (5.39) | 6.86 (5.48) | 7.29 (5.97)

21. Other Pre Specified Outcome: Depression
Description: Assessed using the Patient Health Questionnaire (PHQ-9). This instrument aims to help the diagnosis of depression through the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV), and to determine the severity of the disorder. It is made up of 9 items that refer to the last two weeks. The score ranges between 0 and 27. We only determined it during the washout period (neither early nor late conditions).
  0-4: no depression 5-9: mild depression 10-14: moderate depression 15-19: moderate-severe depression 20-27: severe depression
  Explanation:
  0-4: no depression 5-9: mild depression 10-14: moderate depression 15-19: moderate-severe depression 20-27: severe depression The higher the score, the more harmful
Time Frame: During the week of washout
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Early OGTT, Then Late OGTT in MTNR1B CC | Early OGTT, Then Late OGTT in MTNR1B CG | Early OGTT, Then Late OGTT in MTNR1B GG | Late OGTT, Then Early OGTT in MTNR1B CC | Late OGTT, Then Early OGTT in MTNR1B CG | Late OGTT, Then Early OGTT in MTNR1B GG
Number analyzed (Participants) | 221 | 193 | 36 | 202 | 149 | 44
score | 4.50 (3.89) | 4.61 (4.17) | 4.77 (4.83) | 4.98 (4.52) | 4.57 (3.63) | 5.31 (4.41)

ADVERSE EVENTS:
Time Frame: During 9 days (1 day of intervention-1 week of washout-1 day of intervention), through study completion
Groups:
- Early OGTT (First) in MTNR1B CC; Late OGTT (Second) in MTNR1B CC: Oral glucose tolerance test (OGTT) in homozygous non-carriers (CC) for MTNR1B rs10830963 in Early condition. After a washout period of 1 week, OGTT was performed in Late condition in a randomized cross-over study design.
- Early OGTT (First) in MTNR1B CG: Oral glucose tolerance test (OGTT) in heterozygous (CG) risk allele carriers for MTNR1B rs10830963 in Early condition. After a washout period of 1 week, OGTT was performed in Late condition in a randomized cross-over study design.
- Early OGTT (First) in MTNR1B GG; Late OGTT (Second) in MTNR1B GG: Oral glucose tolerance test (OGTT) in homozygous (GG) risk allele carriers for MTNR1B rs10830963 in Early condition. After a washout period of 1 week, OGTT was performed in Late condition in a randomized cross-over study design.
- Late OGTT (First) in MTNR1B CC; Early OGTT (Second) in MTNR1B CC: Oral glucose tolerance test (OGTT) in homozygous non-carriers (CC) for MTNR1B rs10830963 in Late condition. After a washout period of 1 week, OGTT was performed in Early condition in a randomized cross-over study design.
- Late OGTT (First) in MTNR1B CG; Early OGTT (Second) in MTNR1B CG: Oral glucose tolerance test (OGTT) in heterozygous (CG) risk allele carriers for MTNR1B rs10830963 in Late condition. After a washout period of 1 week, OGTT was performed in Early condition in a randomized cross-over study design.
- Late OGTT (First) in MTNR1B GG; Early OGTT (Second) in MTNR1B GG: Oral glucose tolerance test (OGTT) in homozygous (GG) risk allele carriers for MTNR1B rs10830963 in Late condition. After a washout period of 1 week, OGTT was performed in Early condition in a randomized cross-over study design.
- Late OGTT (Second) in MTNR1B CG: Oral glucose tolerance test (OGTT) in heterozygous (CG) risk allele carriers for MTNR1B rs10830963 in Early condition. After a washout period of 1 week, OGTT was performed in Late condition in a
Arm/Group | Early OGTT (First) in MTNR1B CC | Early OGTT (First) in MTNR1B CG | Early OGTT (First) in MTNR1B GG | Late OGTT (First) in MTNR1B CC | Late OGTT (First) in MTNR1B CG | Late OGTT (First) in MTNR1B GG | Late OGTT (Second) in MTNR1B CC | Late OGTT (Second) in MTNR1B CG | Late OGTT (Second) in MTNR1B GG | Early OGTT (Second) in MTNR1B CC | Early OGTT (Second) in MTNR1B CG | Early OGTT (Second) in MTNR1B GG
All-Cause Mortality (participants affected / at risk) | 0/221 | 0/193 | 0/36 | 0/202 | 0/149 | 0/44 | 0/221 | 0/193 | 0/36 | 0/202 | 0/149 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/221 | 0/193 | 0/36 | 0/202 | 0/149 | 0/44 | 0/221 | 0/193 | 0/36 | 0/202 | 0/149 | 0/44
Other Adverse Events (participants affected / at risk) | 0/221 | 0/193 | 0/36 | 0/202 | 0/149 | 0/44 | 0/221 | 0/193 | 0/36 | 0/202 | 0/149 | 0/44

LIMITATIONS AND CAVEATS:
* Typically, the Participant Flow list Arms/Groups "per sequence" (i.e., "MTNR1B CC Early OGTT first, then Late OGTT", MTNR1B CC Late OGTT first, then Early OGTT", etc.). However, as shown (Diabetes Care, PUBMED: 35015083), the study was conducted to compare the conditions of "early" and "late", within each genotyping-group without considering the order.
* The individual's genotypes were not known until the end of the study, then we could not assign the groups until we finished the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT03036592/Prot_002.pdf
  • Statistical Analysis Plan (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT03036592/SAP_003.pdf
  • Informed Consent Form (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT03036592/ICF_004.pdf